CLINICAL TRIAL: NCT01070303
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of the Human Anti-TNF Monoclonal Antibody Adalimumab for the Maintenance of Clinical Remission in Subjects With Crohn's Disease, Open Label Extension
Brief Title: Remission in Subjects With Crohn's Disease, Open Label Extension
Acronym: CLASSICII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Anne Camez, Medical Director, Abbott
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-433 Open Label
Record Dates: First submitted 2010-02-16; First posted 2010-02-18 (Estimated); Results first posted 2010-05-07 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Crohn's Disease
Keywords: HUMIRA; adalimumab; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab 40 mg every other week or every week (Experimental)
  Interventions: Biological: Adalimumab 40 mg eow or ew

INTERVENTIONS:
Biological: Adalimumab 40 mg eow or ew — Adalimumab 40 mg by subcutaneous injection every other week or every week
  Other Names: Adalimumab; Humira

SUMMARY:
The objectives were: (1) To demonstrate the efficacy of adalimumab in the long-term maintenance of clinical remission in participants with Crohn's disease; and (2) To delineate the long-term safety of adalimumab when administered to participants with Crohn's disease.

DETAILED DESCRIPTION:
Study M02-433 was designed to evaluate the efficacy and safety of adalimumab in the maintenance of clinical remission in patients with Crohn's disease (CD). The study consisted of 2 phases: 1. a 1-year phase (Week 0 to Week 56) (NCT00055497) that consisted of a randomized, double-blind, placebo-controlled portion with a concomitant open label (OL) portion, and 2. a long-term open-label extension (OLE) phase (NCT01070303) that lasted 264 additional weeks (Week 56 to Week 320).

Participants who completed the lead-in study NCT00055523, were eligible to participate in the rollover study, NCT00055497. 176 participants were documented as having completed Year 1 (NCT00055497); however, 177 participants were still receiving study drug and were evaluated at Week 56 of NCT00055497; these participants are included in the OLE data (NCT01070303).

At Week 4 of NCT00055497, participants who demonstrated clinical remission (defined as a Crohn's Disease Activity Index [CDAI] score <150 points) at Baseline of NCT00055497 and who remained in clinical remission at Week 4 ("Remitters") were randomized to receive 1 of 3 blinded treatments: placebo, adalimumab 40 mg every other week (eow), or adalimumab 40 mg every week (ew). Participants who did not demonstrate clinical remission at Baseline of NCT00055497 or who were no longer in clinical remission at Week 4 of NCT00055497 ("Non-remitters") were assigned to receive OL adalimumab 40 mg eow. All study drug (placebo and active) was administered by subcutaneous (SC) injection.

At any time during Study NCT00055497, a participant receiving blinded study drug who developed a disease flare could be switched to OL adalimumab 40 mg eow. A participant receiving OL adalimumab 40 mg SC eow who developed a flare or was a non-responders could have had his/her dose increased to 40 mg SC ew.

After 1 year (Week 56 of NCT00055497), patients who were still participating could continue in the OLE phase (NCT01070303). Participants who were receiving blinded study drug were switched to OL adalimumab 40 mg SC eow, and participants who were receiving OL study drug continued on their previous OL adalimumab dose (adalimumab 40 mg SC eow or ew).

Data are summarized for Remitters and Non-remitters, with the exception of data for primary reason for noncompletion. Summaries of primary reason for noncompletion were available only for all participants, not for Remitters and Non-remitters. Data are reported for Weeks 104, 152, 212, and 260 of Study M02-433, starting from Week 0 of NCT00055497; these weeks correspond to 1, 2, 3, and 4 years of participation in NCT01070303. Change from Baseline results (clinical response 70, clinical response 100, Inflammatory Bowel Disease Questionnaire, and fistula remission) are calculated from Baseline of the lead-in study (NCT00055523). Results on each assessment at each measurement time point are presented as individual outcome measures because different numbers of participants were evaluated at each time point (as observed analysis).

ELIGIBILITY:
Inclusion Criteria:

* Participant had completed the Year 1 of Study M02-433 (NCT00055497)
* Diagnosis of Crohn's disease
* Willing and able to give informed consent

Exclusion Criteria:

* Diagnosis of ulcerative colitis
* Pregnancy or breastfeeding
* Previous use of infliximab or other anti-TNF (tumor necrosing factor) antagonists
* Previous history of active tuberculosis or listeria infection
* Previous history of cancer other than successfully treated skin cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2002-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Camez, MD, Study Director — Abbott
Locations (43):
- United States (43):
  - Gastroenterology Associates of the East Bay, Berkeley, California
  - Long Beach Gastroenterology Assoc., Long Beach, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Gastroenterology Assoc. of Fairfield Co., Bridgeport, Connecticut
  - Cleveland Clinic Florida, Weston, Florida
  - Wake Research Associates, Weston, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Assoc., Atlanta, Georgia
  - Southeastern Digestive & Liver Disease, Savannah, Georgia
  - Northwest Gastroenterologists, S.C., Arlington Heights, Illinois
  - University of Chicago, Chicago, Illinois
  - Drug Research Services, Inc., Metairie, Louisiana
  - LSU School of Medicine, New Orleans, Louisiana
  - Digestive Disorders Associates, Annapolis, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clinical Pharmacology Study Group, Worchester, Massachusetts
  - Mayo Clinic and Mayo Foundation, Rochester, Minnesota
  - Gastroenterology and Hepatology, Kansas City, Missouri
  - Glenn Gordon, MD, Mexico, Missouri
  - Deaconess Billings Clinic Research Division, Billings, Montana
  - Gastroenterology Specialties, P.C., Lincoln, Nebraska
  - Long Island Clinical Research Associates, Great Neck, New York
  - NY Center for Clinical Research, Lake Success, New York
  - New York Presbyterian Hospital, New York, New York
  - Daniel Present, New York, New York
  - Rochester Institute for Digestive Diseases, Rochester, New York
  - UNC School of Medicine, Chapel Hill, North Carolina
  - Charlotte Gastroenterology and Hepatology, Charlotte, North Carolina
  - Carolina Research Associates, Charlotte, North Carolina
  - Digestive Health Specialists, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Oklahoma Foundation for Digestive Disease, Oklahoma City, Oklahoma
  - Research Solutions, Tulsa, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Peter Molloy, MD, Pittsburgh, Pennsylvania
  - Diseases of the Digestive System, Chattanooga, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Northwest Gastroenterology, Bellevue, Washington
  - Inland Empire Gastroenterology, Spokane, Washington
  - Tacoma Digestive Disease Center, Tacoma, Washington
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Ryan C, Sobell JM, Leonardi CL, Lynde CW, Karunaratne M, Valdecantos WC, Hendrickson BA. Safety of Adalimumab Dosed Every Week and Every Other Week: Focus on Patients with Hidradenitis Suppurativa or Psoriasis. Am J Clin Dermatol. 2018 Jun;19(3):437-447. doi: 10.1007/s40257-017-0341-6. PMID 29380251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were still receiving study drug and were evaluated at Week 56 of Study M02-433 (NCT00055497) are included in the open-label extension (OLE) (NCT01070303). Participants entered NCT00055497 from a lead-in adalimumab induction therapy study (NCT00055523).
Pre-assignment Details: Clinical remission = CDAI <150. At Week 4 of NCT00055497, "remitters" (participants in clinical remission at Week 0 and Week 4 of NCT00055497) were randomized to double blind (DB) therapy and "non-remitters" (participants not in clinical remission at Week 0 or no longer in clinical remission at Week 4) were assigned to open-label (OL) adalimumab.
Groups:
- All Participants in Open-Label Extension of Study M02-433: Participants who were still receiving study drug and were evaluated at Week 56 of NCT00055497 could continue into the OLE. In the OLE, participants who received double-blind study drug (adalimumab 40 mg) during the DB portion were started on adalimumab 40 mg every other week (eow). Participants who received OL adalimumab 40 mg during the DB portion continued the dose they were receiving. Any participant who was receiving 40 mg adalimumab eow during the OLE and who experienced a disease flare (recurrence of active disease) could change to 40 mg adalimumab weekly. 176 participants were documented as completing Year 1 of the study; however, efficacy data were recorded for 177 participants at Week 56, and those participants are included in the OLE. Safety data are summarized for all participants (N = 276) who entered the study (NCT00055497).
Period: Overall Study
Arm/Group | All Participants in Open-Label Extension of Study M02-433
Started | 177
Completed | 88
Not Completed | 89
Not completed — Adverse Event | 39
Not completed — Withdrawal by Subject | 20
Not completed — Lost to Follow-up | 9
Not completed — Protocol Violation | 0
Not completed — Lack of Efficacy | 2
Not completed — Administrative Reason | 1
Not completed — Other | 18

BASELINE CHARACTERISTICS:
Groups:
- Remitters: Adalimumab 40 mg by subcutaneous injection every other week or every week. Baseline remitters were subjects who demonstrated clinical remission (CDAI score < 150 points) at Week 0 of NCT00055497 and remained in clinical remission at Week 4 of NCT00055497.
- Non-Remitters: Adalimumab 40 mg by subcutaneous injection every other week or every week. Baseline non-remitters were subjects who did not demonstrate clinical remission at Week 0 of NCT00055497, or who were no longer in remission at Week 4 of NCT00055497.
- Total: Total of all reporting groups
Arm/Group | Remitters | Non-Remitters | Total
Number analyzed (Participants) | 45 | 132 | 177
Age Continuous [Mean (Standard Deviation); unit: years] | 35.5 (10.88) | 38.9 (12.53) | 38.1 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 60 | 86
  Male | 19 | 72 | 91
Region of Enrollment [Number; unit: participants]
  United States | 45 | 132 | 177

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Clinical Remission (Crohn's Disease Activity Index[CDAI] <150 Points) at Week 104 of Study M02-433 (Starting From Week 0 of NCT00055497) (Through 1 Year of Participation in NCT01070303).
Description: Clinical remission is defined as CDAI score <150. CDAI evaluates 8 Crohn's-related variables during a 1-week assessment period, yielding a composite score >/= 0 and without upper limit. The range of scores during Study NCT01070303 was 0 to 464. A lower score indicates less severe Crohn's disease activity.
Time Frame: Week 104
Population: The analysis population is observed cases, that is, all participants who had CDAI evaluation at Week 104 are included.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 34 | 103
Participants | 29 | 71

2. Secondary Outcome: Number of Participants Achieving Clinical Remission (CDAI < 150 Points) at Week 152 (Through 2 Years of Participation in NCT01070303).
Description: as for outcome 1
Time Frame: Week 152
Population: The analysis population is observed cases, that is, all participants who had CDAI evaluation at Week 152 are included.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 30 | 87
Participants | 26 | 62

3. Secondary Outcome: Number of Participants Achieving Clinical Remission (CDAI < 150 Points) at Week 212 (Through 3 Years of Participation in NCT01070303).
Description: as for outcome 1
Time Frame: Week 212
Population: Observed cases, that is, all participants who participating at Week 212 and had a CDAI measurement at that time point were included.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 25 | 69
Participants | 21 | 45

4. Secondary Outcome: Number of Participants Achieving Clinical Remission (CDAI < 150 Points) at Week 260 (4 Years of Participation in NCT01070303).
Description: as for outcome 1
Time Frame: Week 260
Population: The analysis population is observed cases, that is, all participants who had CDAI evaluation at Week 260 of Study NCT00055497 are included.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 10 | 27
Participants | 8 | 21

5. Secondary Outcome: Number of Participants Achieving CR-100 at Week 104 (1 Year of Participation in NCT01070303)
Description: A CR-100 is a decrease from Baseline of lead-in study (NCT00055523) in CDAI score of 100 or more points, indicating significant improvement in disease severity. CDAI evaluates 8 Crohn's-related variables during a 1-week assessment period, yielding a composite score >/= 0 and without upper limit. The range of scores during Study NCT01070303 was 0 to 464. Scores at Baseline of the lead-in study (NCT00055523), which were used to calculate clinical response, ranged from 201 to 450. A lower score indicates less severe Crohn's disease activity.
Time Frame: From Baseline of lead-in study to Week 104
Population: The analysis population is observed cases, that is, all participants who had CDAI evaluation at Week 104 of Study NCT00055497 are included.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 34 | 103
Participants | 28 | 87

6. Secondary Outcome: Number of Participants Achieving CR-100 at Week 152 (2 Years of Participation in NCT01070303)
Description: A CR-100 is a decrease from Baseline of lead-in study (NCT00055523) in CDAI score of 100 or more points, indicating a significant improvement in disease severity. CDAI evaluates 8 Crohn's-related variables during a 1-week assessment period, yielding a composite score >/= 0 and without upper limit. The range of scores during Study NCT01070303 was 0 to 464. Scores at Baseline of the lead-in study (NCT00055523), which were used to calculate clinical response, ranged from 201 to 450. A lower score indicates less severe Crohn's disease activity.
Time Frame: From Baseline of lead-in study to Week 152
Population: The analysis population is observed cases, that is, all participants who had CDAI evaluation at Week 152 are included.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 30 | 87
Participants | 28 | 74

7. Secondary Outcome: Number of Participants Achieving CR-100 at Week 212 (3 Years of Participation in NCT01070303)
Description: as for outcome 6
Time Frame: From Baseline of lead-in study to Week 212
Population: The analysis population is observed cases, that is, all participants who had CDAI evaluation at Week 212
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 25 | 69
Participants | 23 | 58

8. Secondary Outcome: Number of Participants Achieving CR-100 at Week 260 (4 Years of Participation in NCT01070303)
Description: as for outcome 5
Time Frame: From Baseline of lead-in study to Week 260
Population: The analysis population is observed cases, that is, all participants who had CDAI evaluation at Week 260 are included.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 10 | 27
Participants | 8 | 27

9. Secondary Outcome: Number of Participants Achieving CR-70 at Week 104 (1 Year of Participation in NCT01070303)
Description: A CR-70 is a decrease from Baseline of lead-in study (NCT00055523) in CDAI score of 70 or more points, indicating a significant improvement in disease severity. CDAI evaluates 8 Crohn's-related variables during a 1-week assessment period, yielding a composite score >/= 0 and without upper limit. The range of scores during Study NCT01070303 was 0 to 464. Scores at Baseline of the lead-in study (NCT00055523), which were used to calculate clinical response, ranged from 201 to 450. A lower score indicates less severe Crohn's disease activity.
Time Frame: Week 104
Population: The analysis population is observed cases, that is, all participants who had CDAI evaluation at Week 104 .
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 34 | 103
Participants | 31 | 92

10. Secondary Outcome: Number of Participants Achieving CR-70 at Week 152 (2 Years of Participation in NCT01070303)
Description: as for outcome 9
Time Frame: From Baseline of lead-in Study to Week 152
Population: The analysis population is observed cases, that is, all participants who CDAI evaluation at Week 152 are included.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 30 | 87
Participants | 30 | 77

11. Secondary Outcome: Number of Participants Achieving CR-70 at Week 212 (3 Years of Participation in NCT01070303)
Description: CR-70 is a decrease from Baseline of lead-in study (NCT00055523) in CDAI score of 70 or more points, indicating a significant improvement in disease severity. CDAI evaluates 8 Crohn's-related variables during a 1-week assessment period, yielding a composite score >/= 0 and without upper limit. The range of scores during Study NCT01070303 was 0 to 464. Scores at Baseline of the lead-in study (NCT00055523), which were used to calculate clinical response, ranged from 201 to 450. A lower score indicates less severe Crohn's disease activity.
Time Frame: From Baseline of lead-in study to Week 212
Population: The analysis population is observed cases, that is, all participants who had CDAI evaluation Week 212 are included.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 25 | 69
Participants | 24 | 63

12. Secondary Outcome: Number of Participants Achieving CR-70 at Week 260 (4 Years of Participation in NCT01070303)
Description: as for outcome 9
Time Frame: From Baseline of lead-in study to Week 260
Population: The analysis population is observed cases, that is, all participants who had CDAI evaluation at Week 260 are included.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 10 | 27
Participants | 10 | 27

13. Secondary Outcome: Number of Participants Achieving Steroid-free Clinical Remission at Week 104 (1 Year of Participation in NCT01070303)
Description: Among participants who were taking systemic corticosteroids at Baseline of the lead-in study (NCT00055523), steroid-free remission was achieved if the participant stopped taking corticosteroids before the visit and had a CDAI score < 150 points at that visit.
Time Frame: From Baseline of lead-in study to Week 104
Population: The analysis population was observed cases, that is, all participants who were taking systemic corticosteroids at Baseline of NCT00055523 and who had CDAI evaluation and documentation of concomitant corticosteroid use (yes or no) at Week 104.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 18 | 31
Participants | 8 | 12

14. Secondary Outcome: Number of Achieving Steroid-free Clinical Remission at Week 152 (2 Years of Participation in NCT01070303)
Description: as for outcome 13
Time Frame: From Baseline of lead-in study to Week 152
Population: The analysis population was observed cases, that is, all participants who were taking systemic corticosteroids at Baseline of NCT00055523 and who had CDAI evaluation and documentation of concomitant corticosteroid use (yes or no) at Week 152.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 18 | 30
Participants | 8 | 14

15. Secondary Outcome: Number of Participants Achieving Steroid-free Clinical Remission at Week 212 (3 Years of Participation in NCT01070303)
Description: as for outcome 13
Time Frame: From Baseline of lead-in study to Week 212
Population: The analysis population was observed cases, that is, all participants who were taking systemic corticosteroids at Baseline of NCT00055523 and who had CDAI evaluation and documentation of concomitant corticosteroid use (yes or no) at Week 212.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 14 | 23
Participants | 5 | 10

16. Secondary Outcome: Number of Participants Achieving Steroid-free Clinical Remission at Week 260 (4 Years of Participation in NCT01070303)
Description: as for outcome 13
Time Frame: From Baseline of lead-in study to Week 260
Population: The analysis population was observed cases, that is, all participants who were taking systemic corticosteroids at Baseline of NCT00055523 and who had CDAI evaluation and documentation of concomitant corticosteroid use (yes or no) at Week 260.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 6 | 12
Participants | 2 | 4

17. Secondary Outcome: Number of Participants Achieving Steroid-free CR-100 at Week 104 (1 Year of Participation in NCT01070303)
Description: Among participants who were taking systemic corticosteroids at Baseline of the lead-in study (NCT00055523), steroid-free CR-100 was achieved if the participant stopped taking steroids before the visit and had a decrease from Baseline in CDAI score of 100 or more points at that visit.
Time Frame: From Baseline of lead-in study to Week 104
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 18 | 31
Participants | 9 | 15

18. Secondary Outcome: Number of Participants Achieving Steroid-free CR-100 at Week 152 (2 Years of Participation in NCT01070303)
Description: as for outcome 17
Time Frame: From Baseline of lead-in study to Week 152
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 18 | 30
Participants | 9 | 15

19. Secondary Outcome: Number of Participants Achieving Steroid-free CR-100 at Week 212 (3 Years of Participation in NCT01070303)
Description: as for outcome 17
Time Frame: From Baseline of lead-in study to Week 212
Population: as for outcome 15
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 14 | 23
Participants | 6 | 12

20. Secondary Outcome: Number of Participants Achieving Steroid-free CR-100 at Week 260 (4 Years of Participation in NCT01070303)
Description: as for outcome 17
Time Frame: From Baseline of lead-in study to Week 260
Population: as for outcome 16
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 6 | 12
Participants | 2 | 5

21. Secondary Outcome: Changes in Inflammatory Bowel Disease Questionnaire (IBDQ) Scores
Description: IBDQ is a validated disease-specific instrument that assesses the impact of IBD on patient quality of life during a 2-week recall period. It has 32 questions about bowel function and related symptoms, and their social and emotional impact. For each question, participants selected 1 of 7 responses, where 1=poor quality of life (e.g., feeling of fatigue "all of the time") and 7=good quality on the item (e.g., feeling of fatigue "none of the time"). IBDQ scores range from 32 to 224. Higher scores indicate better quality of life, and increases in IBDQ indicate improved overall quality of life.
Time Frame: Change from Baseline of lead-in study at Weeks 104, 152, 200, and 248
Population: The analysis population is observed cases, that is, all participants who had an IBDQ score at the visit time point.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Change From Baseline-Week 104; Change From Baseline-Week 152; Change From Baseline-Week 200; Change From Baseline-Week 248: The last non-missing measure collected on or before the first dose of study drug in the lead-in study, NCT00055523, was used as Baseline to determine efficacy changes. Only participants who had Baseline and post Baseline visits were included in the analyses.
Arm/Group | Change From Baseline-Week 104 | Change From Baseline-Week 152 | Change From Baseline-Week 200 | Change From Baseline-Week 248
Number analyzed (Participants) | 142 | 114 | 99 | 69
Scores on a scale | 42.4 (36.27) | 47.9 (33.70) | 51.0 (32.77) | 51.7 (32.67)

22. Secondary Outcome: Number of Participants Achieving Fistula Remission at Week 104 (1 Year of Participation in NCT01070303)
Description: A count of the number of cutaneous fistulas draining upon gentle compression was performed at Baseline of the lead-in study (NCT00055523) and at study visits. Among participants with draining fistulas at Baseline of NCT00055523, a participant was considered to have achieved fistula remission at a study visit if the participant had no draining cutaneous fistulas at that visit.
Time Frame: From Baseline of lead-in study to Week 104
Population: The analysis population was observed cases, that is, all participants who draining fistulas at Baseline of NCT00055523 and who had data on draining fistulas(yes or no) at Week 104.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 3 | 15
Participants | 1 | 11

23. Secondary Outcome: Number of Participants Achieving Fistula Remission at Week 152 (2 Years of Participation in NCT01070303)
Description: as for outcome 22
Time Frame: From Baseline of lead-in study to Week 152
Population: The analysis population was observed cases, that is, all participants who draining fistulas at Baseline of NCT00055523 and who had data on draining fistulas(yes or no) at Week 152.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 3 | 14
Participants | 2 | 11

24. Secondary Outcome: Number of Participants Achieving Fistula Remission at Week 212 (3 Years of Participation in NCT01070303)
Description: as for outcome 22
Time Frame: From Baseline of lead-in study to Week 212
Population: The analysis population was observed cases, that is, all participants who draining fistulas at Baseline of NCT00055523 and who had data on draining fistulas(yes or no) at Week 212.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 3 | 11
Participants | 1 | 10

25. Secondary Outcome: Number of Participants Achieving Fistula Remission at Week 260 (Years of Participation in NCT01070303)
Description: as for outcome 22
Time Frame: From Baseline of lead-in study to Week 260
Population: The analysis population was observed cases, that is, all participants who draining fistulas at Baseline of NCT00055523 and who had data on draining fistulas(yes or no) at Week 260.
Measure: Number; unit: Participants
Arm/Group | Remitters | Non-Remitters
Number analyzed (Participants) | 2 | 7
Participants | 2 | 6

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs), defined as AEs beginning on or after first dose of adalimumab (in NCT00055523, NCT00055497, or NCT01070303) are reported. Treatment-emergent AEs were recorded up to 70 days after last dose of adalimumab.
Description: Adverse events are reported for all participants who entered the study (NCT00055497), N=276. These 276 participants include the 177 participants who continued into the open-label extension (NCT01070303).
Arm/Group | Remitters | Non-Remitters
Serious Adverse Events (participants affected / at risk) | 6/55 | 69/221
Other Adverse Events (participants affected / at risk) | 50/55 | 207/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remitters (N=55) | Non-Remitters (N=221)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colonic stenosis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 17
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Ileal stenosis (Gastrointestinal disorders) | 1 | 3
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 8
Small intestinal stenosis (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 2
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 1
Nocardiosis (Infections and infestations) | 0 | 1
Parvovirus infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 2
Retroperitoneal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Obesity (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Langerhans' cell granulomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Optic neuritis (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remitters (N=55) | Non-Remitters (N=221)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 11
Abdominal discomfort (Gastrointestinal disorders) | 3 | 5
Abdominal distension (Gastrointestinal disorders) | 3 | 23
Abdominal pain (Gastrointestinal disorders) | 12 | 42
Abdominal pain upper (Gastrointestinal disorders) | 3 | 10
Abdominal tenderness (Gastrointestinal disorders) | 3 | 23
Anal fistula (Gastrointestinal disorders) | 1 | 17
Constipation (Gastrointestinal disorders) | 5 | 17
Crohn's disease (Gastrointestinal disorders) | 23 | 70
Diarrhoea (Gastrointestinal disorders) | 8 | 36
Dyspepsia (Gastrointestinal disorders) | 4 | 23
Flatulence (Gastrointestinal disorders) | 2 | 17
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 22
Nausea (Gastrointestinal disorders) | 8 | 51
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 19
Tooth impacted (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 4 | 28
Chest pain (General disorders) | 2 | 14
Fatigue (General disorders) | 6 | 26
Influenza like illness (General disorders) | 2 | 18
Injection site irritation (General disorders) | 9 | 21
Injection site pain (General disorders) | 3 | 12
Injection site reaction (General disorders) | 2 | 22
Pain (General disorders) | 0 | 12
Pyrexia (General disorders) | 5 | 33
Seasonal allergy (Immune system disorders) | 3 | 2
Bronchitis (Infections and infestations) | 3 | 15
Fungal infection (Infections and infestations) | 1 | 12
Gastroenteritis (Infections and infestations) | 1 | 13
Influenza (Infections and infestations) | 8 | 28
Nasopharyngitis (Infections and infestations) | 15 | 50
Pharyngitis streptococcal (Infections and infestations) | 3 | 4
Respiratory tract infection viral (Infections and infestations) | 3 | 3
Sinusitis (Infections and infestations) | 6 | 34
Tooth abscess (Infections and infestations) | 3 | 8
Upper respiratory tract infection (Infections and infestations) | 8 | 30
Urinary tract infection (Infections and infestations) | 4 | 24
Viral infection (Infections and infestations) | 5 | 12
Excoriation (Injury, poisoning and procedural complications) | 3 | 5
Antinuclear antibody positive (Investigations) | 3 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 43
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 31
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 13
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 19
Dizziness (Nervous system disorders) | 5 | 12
Headache (Nervous system disorders) | 8 | 47
Anxiety (Psychiatric disorders) | 5 | 13
Depression (Psychiatric disorders) | 4 | 16
Insomnia (Psychiatric disorders) | 4 | 26
Haematuria (Renal and urinary disorders) | 3 | 10
Nephrolithiasis (Renal and urinary disorders) | 2 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 17
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 12
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Acne (Skin and subcutaneous tissue disorders) | 2 | 12
Eczema (Skin and subcutaneous tissue disorders) | 3 | 14
Erythema (Skin and subcutaneous tissue disorders) | 7 | 9
Pruritis (Skin and subcutaneous tissue disorders) | 5 | 10
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 7
Rash (Skin and subcutaneous tissue disorders) | 8 | 32
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 | 4
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 | 2
Hypertension (Vascular disorders) | 1 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.